CLINICAL TRIAL: NCT03247738
Title: Platelet Inhibition With CANgrelor and Crushed TICagrelor in STEMI Patients Undergoing Primary Percutaneous Coronary Intervention: The CANTIC Study
Brief Title: Platelet Inhibition With Cangrelor and Crushed Ticagrelor in STEMI
Acronym: CANTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIS CHI001 WIRB
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Results first posted 2020-02-06 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: ST Segment Elevation Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: ticagrelor; cangrelor
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — cangrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cangrelor (Experimental): Cangrelor will be administered as 30 μg/kg bolus followed by 4 μg/kg/min infusion for 2 hours
  Interventions: Drug: Cangrelor
- Placebo (Placebo Comparator): Normal saline bolus and infusion for 2 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cangrelor — Patients will be randomly assigned 1:1 to receive either cangrelor or matching placebo. The bolus will be administered at the same time of a 180 mg crushed ticagrelor loading dose and infusion will be continued for 2 h.
  Other Names: Kangreal
  Arms: Cangrelor
Other: Placebo — Patients will be randomly assigned 1:1 to receive either cangrelor or matching placebo. The bolus will be administered at the same time of a 180 mg crushed ticagrelor loading dose and infusion will be continued for 2 h.
  Arms: Placebo

SUMMARY:
In STEMI patients undergoing PPCI there is a delayed onset of action of oral P2Y12 receptor inhibitors, including prasugrel and ticagrelor. Crushing prasugrel and ticagrelor improves their PK and PD profiles as it favors drug absorption and onset of antiplatelet effects and because of this, it is commonly used in STEMI patients undergoing PPCI. However, despite the use of crushed tablets, up to one-third of patients may still have high on-treatment platelet reactivity (HPR) within the first 2 hours after loading dose (LD) administration of these oral agents. Cangrelor is a potent intravenous P2Y12 receptor inhibitor with rapid onset and offset of action associated with a greater reduction in ischemic events compared with clopidogrel in P2Y12 receptor naïve patients undergoing PCI. To date most studies have explored cangrelor in the setting of PCI subjects treated with clopidogrel. The PD effects of cangrelor in STEMI patients undergoing PPCI treated with a newer generation P2Y12 receptor inhibitor and how this compares with a crushed formulation of the oral drug is unexplored. The aim of this prospective randomized study is to investigate the PD effects of cangrelor in STEMI patients undergoing PPCI treated with crushed ticagrelor.

DETAILED DESCRIPTION:
In STEMI patients undergoing PPCI there is a delayed onset of action of oral P2Y12 receptor inhibitors, including prasugrel and ticagrelor, which require more than 2 hours to exert their full antiplatelet effects, and thus exposing these high-risk patients to an increased risk of early thrombotic complications. The mechanism of this delayed onset of antiplatelet effect is likely multifactorial due to the presence in the setting of STEMI of specific conditions that translate into delayed drug absorption which in turn affect the pharmacokinetic (PK) and pharmacodynamic (PD) profiles of oral P2Y12 receptor inhibitors. Crushing prasugrel and ticagrelor improves their PK and PD profiles as it favors drug absorption and onset of antiplatelet effects and because of this, it is commonly used in STEMI patients undergoing PPCI. However, despite the use of crushed tablets, up to one-third of patients may still have high on-treatment platelet reactivity (HPR) within the first 2 hours after loading dose (LD) administration of these oral agents. Cangrelor is a potent intravenous P2Y12 receptor inhibitor with rapid onset and offset of action associated with a greater reduction in ischemic events compared with clopidogrel in P2Y12 receptor naïve patients undergoing PCI. To date most studies have explored cangrelor in the setting of PCI subjects treated with clopidogrel and the clinical profile of cangrelor among patients treated with prasugrel or ticagrelor is currently unknown. This is noteworthy because ACS patients, in particular STEMI undergoing PPCI, are commonly treated with either prasugrel or ticagrelor. PD investigations conducted in vitro or ex vivo in stable patients have shown cangrelor to be associated with enhanced platelet inhibition compared with that induced by prasugrel and ticagrelor. However, the PD effects of cangrelor in STEMI patients undergoing PPCI treated with a newer generation P2Y12 receptor inhibitor and how this compares with a crushed formulation of the oral drug is unexplored. The aim of this prospective randomized study is to investigate the PD effects of cangrelor in STEMI patients undergoing PPCI treated with crushed ticagrelor.

ELIGIBILITY:
Inclusion criteria:

* Patients with STEMI undergoing primary PPCI
* Age > 18 years old

Exclusion criteria:

* Inability to provide written informed consent
* Known history of prior intracranial bleeding
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) in the prior 10 days
* Known allergies to aspirin, ticagrelor or cangrelor
* On treatment with oral anticoagulant
* Treatment with glycoprotein IIb/IIIa inhibitors
* Fibrinolytics within 24 hours
* Active bleeding
* High risk of bleeding
* Known platelet count <80x106/mL
* Known hemoglobin <10 g/dL
* Intubated patients (prior to randomization)
* Known creatinine clearance <30 mL/minute or on hemodialysis.
* Known severe hepatic dysfunction
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luker J, Kuhr K, Sultan A, Nolker G, Omran H, Willems S, Andrie R, Schrickel JW, Winter S, Vollmann D, Tilz RR, Jobs A, Heeger CH, Metzner A, Meyer S, Mischke K, Napp A, Fahrig A, Steinhauser S, Brachmann J, Baldus S, Mahajan R, Sanders P, Steven D. Internal Versus External Electrical Cardioversion of Atrial Arrhythmia in Patients With Implantable Cardioverter-Defibrillator: A Randomized Clinical Trial. Circulation. 2019 Sep 24;140(13):1061-1069. doi: 10.1161/CIRCULATIONAHA.119.041320. Epub 2019 Aug 30. PMID 31466479
- [Derived] Franchi F, Rollini F, Rivas A, Wali M, Briceno M, Agarwal M, Shaikh Z, Nawaz A, Silva G, Been L, Smairat R, Kaufman M, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Bass TA, Angiolillo DJ. Platelet Inhibition With Cangrelor and Crushed Ticagrelor in Patients With ST-Segment-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention. Circulation. 2019 Apr 2;139(14):1661-1670. doi: 10.1161/CIRCULATIONAHA.118.038317. PMID 30630341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 10, 2017 and July 17, 2018, there were a total of 99 STEMI patients with intent to undergo P-PCI that presented to our Institution, of whom 69 provided their written informed consent to participate in the study.
Pre-assignment Details: 19 patients were not randomized because PCI was not performed or had newly identified exclusion criteria
Period: Overall Study
Arm/Group | Cangrelor | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cangrelor | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11) | 60 (10) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 20 | 16 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Radial access [Count of Participants; unit: Participants] | 20 | 20 | 40
Use of glycoprotein IIb/IIIa inhibitors [Count of Participants; unit: Participants] | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured by VerifyNow PRU
Description: Platelet reactivity at 30 minutes after starting cangrelor or placebo assessed by VerifyNow PRU and reported as P2Y12 Reaction Units (PRU)
Time Frame: 30 minutes
Population: The analyzed patients included all patients with pharmacodynamic data and without a major protocol deviation thought to affect the pharmacodynamic effects of ticagrelor or cangrelor.
Measure: Least Squares Mean (95% Confidence Interval); unit: P2Y12 reaction units (PRU)
Arm/Group | Cangrelor | Placebo
Number analyzed (Participants) | 22 | 22
P2Y12 reaction units (PRU) | 63 [32 to 93] | 214 [183 to 245]
Statistical Analysis 1: Comparison: Cangrelor vs Placebo; Test type: Superiority — The primary end point of our study was the comparison of platelet reactivity measured by VerifyNow PRU between cangrelor and placebo at 30 minutes after drugs were administered at the start of PCI. Assuming a common standard deviation of 70 PRU, a sample size of 20 patients per group would allow detection of a 70 PRU difference between groups with 85% power and a two-sided α = 0.05. Considering the 2 arms and a possible 25% rate of invalid PD results we planned to randomize up to 50 patients; p < 0.001, ANCOVA; the baseline value of platelet reactivity used as a covariate; Mean Difference (Net) = 152, 95% CI 2-sided [108 to 195]

2. Secondary Outcome: Platelet Reactivity Measured by Vasodilator-stimulated Phosphoprotein (VASP)
Description: Platelet reactivity at 30 minutes after starting cangrelor or placebo measured by VASP and reported as platelet reactivity index (PRI%). Higher PRI% means higher platelet reactivity.
Time Frame: 30 minutes
Measure: Least Squares Mean (95% Confidence Interval); unit: platelet reactivity index (PRI)
Arm/Group | Cangrelor | Placebo
Number analyzed (Participants) | 22 | 22
platelet reactivity index (PRI) | 29 [18 to 39] | 72 [61 to 82]

ADVERSE EVENTS:
Time Frame: Until time of discharge
Description: The safety population was composed of all patients exposed to at least one dose of study medication (any time from randomization until completion of the study). Any adverse event until time of discharge was recorded.
Arm/Group | Cangrelor | Placebo
All-Cause Mortality (participants affected / at risk) | 1/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 3/25 | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cangrelor (N=25) | Placebo (N=25)
Acute stent thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cangrelor (N=25) | Placebo (N=25)
minor bleeding (Vascular disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03247738/Prot_SAP_000.pdf